CLINICAL TRIAL: NCT00115375
Title: Dose-Ranging Pharmacodynamic Assessment of Platelet Aggregation Inhibition With Clopidogrel in Children of Blalock-Taussig Shunt Age Categories (Neonates and Infants/Toddlers)
Brief Title: Platelet Aggregation Inhibition in Children on Clopidogrel (PICOLO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDY4422
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Congenital Heart Defects; Blood Platelet Disorders
Keywords: THROMBOSIS; PLATELET AGGREGATION; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital; Blood Platelet Disorders; Thrombosis | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel (SR25990)

SUMMARY:
PICOLO is a double blind placebo controlled phase II dose ranging, dose escalating study in patients of Blalock-Taussig age categories (neonates and infants/toddlers), to determine the dose providing inhibition of platelet aggregation similar to adults.

DETAILED DESCRIPTION:
There will be 3 blinded dose groups of 12 patients each (9 active, 3 placebo), central randomization, stratified by age (< 1 month ;1 to 24 months). There will be a comparison of ADP-induced platelet aggregation at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Neonates or infants/toddlers (up to 24 months) at risk for thrombosis (e.g., Blalock-Taussig shunt or any systemic to pulmonary artery shunt, Kawasaki disease, vascular stent or any condition requiring antiplatelet therapy).

Exclusion Criteria:

* Ongoing bleeding or increased risk of bleeding

  * Weight < 2 kg; gestational age < 35 weeks
  * Allergy to drugs
  * Current or planned anticoagulant treatment
  * Unable to receive drug enterically
  * Platelet transfusion < 7days
  * Thrombocytopenia
  * Hepatic or renal failure

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2004-01; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Percent inhibition of maximum extent and rate of aggregation of 5 µM ADP-induced platelet aggregation

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy

REFERENCES:
- [Result] Li JS, Yow E, Berezny KY, Bokesch PM, Takahashi M, Graham TP Jr, Sanders SP, Sidi D, Bonnet D, Ewert P, Jennings LK, Michelson AD; PICOLO Investigators. Dosing of clopidogrel for platelet inhibition in infants and young children: primary results of the Platelet Inhibition in Children On cLOpidogrel (PICOLO) trial. Circulation. 2008 Jan 29;117(4):553-9. doi: 10.1161/CIRCULATIONAHA.107.715821. Epub 2008 Jan 14. PMID 18195173
- [Derived] Pasquali SK, Yow E, Jennings LK, Li JS. Platelet activity associated with concomitant use of clopidogrel and proton pump inhibitors in children with cardiovascular disease. Congenit Heart Dis. 2010 Nov-Dec;5(6):552-5. doi: 10.1111/j.1747-0803.2010.00461.x. PMID 21106014